CLINICAL TRIAL: NCT00566007
Title: Trial on the Effect of Ozone Therapy for Lumbar Herniated Disc With Criteria for Surgery
Brief Title: The Effect of Ozone Therapy for Lumbar Herniated Disc
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: It has proved extremely difficult
Sponsor: Kovacs Foundation (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other); Hospital Negrín (Unknown); Hospital Son Llatzer (Other); Servicio de Salud de las Islas Baleares (Ib-Salut) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FK-R-21
Record Dates: First submitted 2007-11-29; First posted 2007-11-30 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Lumbar Herniated Disc
Keywords: disc herniation; lumbar; ozone therapy
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Diskectomy; Oxygen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Discectomy/micro discectomy
  Interventions: Procedure: Discectomy/ micro discectomy; Drug: Ozone therapy; Drug: Oxygen therapy
- 2 (Active Comparator): Intradiscal ozone infiltration
  Interventions: Drug: Ozone therapy; Drug: Oxygen therapy
- 3 (Active Comparator): Intradiscal oxygen infiltration (control arm)
  Interventions: Drug: Oxygen therapy

INTERVENTIONS:
Procedure: Discectomy/ micro discectomy — Standard discectomy or micro discectomy
  Arms: 1
Drug: Ozone therapy — Infiltration of intradiscal ozone: O3/O2 in a 27 micrograms/ml concentration + foraminal infiltration of O3/O2 + corticoid + anesthetic
  Arms: 1; 2
Drug: Oxygen therapy — Intradiscal oxygen therapy: O3/O2 at a concentration of 0 micrograms/ml (only oxygen) + foraminal infiltration of O2 + corticoid + anesthetic

SUMMARY:
The purpose of this study is to assess the efficacy (vs. placebo) of ozone infiltration and its effectiveness in comparison with micro discectomy in the treatment of lumbar herniated disc with criteria for surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of herniated disc by surgeons from participating hospitals
* Sciatic pain of 5 or more on Visual Analogue Scale
* Pain radiated to appropriate area according to herniated disc
* On waiting list for disc surgery at one of participating hospitals

Exclusion Criteria:

* Inability to fill out questionnaires (VAS, Roland Morris, SF12)
* Calcified or migrated herniated disc
* Herniated disc with indications for laminectomy or arthrodesis
* Clinically relevant partial paralysis
* Simultaneous cervical and dorsal symptomatic herniated discs
* Previous lumbar spine surgery
* Presence of other spinal pathology
* Significant glucose-6-phosphate-dehydrogenase deficit
* Allergy to ozone
* Treatment with oral anticoagulants

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2008-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of infiltration with corticoids+anesthetics+ozone in comparison with corticoids+anesthetics+oxygen (considered placebo for ozone) | 12 months

SECONDARY OUTCOMES:
To evaluate the effectiveness of both types of infiltration (used in primary outcome) in comparison with discectomy/micro discectomy | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Francisco M Kovacs, MD, PhD, Study Chair — Kovacs Foundation, Palma de Mallorca, 07012, Spain; Bernardino Clavo, MD, Study Director — Hospital Negrín, Las Palmas de Gran Canaria, 35010 Spain; Francisco Robaina, MD, Principal Investigator — Hospital Negrín, Las Palmas de Gran Canaria 35010 Spain
Locations (1):
- Hospital Negrín, Las Palmas de Gran Canaria, Canary Islands, Spain

REFERENCES:
- [Background] Andreula CF, Simonetti L, De Santis F, Agati R, Ricci R, Leonardi M. Minimally invasive oxygen-ozone therapy for lumbar disk herniation. AJNR Am J Neuroradiol. 2003 May;24(5):996-1000. PMID 12748111
- [Background] Bonetti M, Fontana A, Cotticelli B, Volta GD, Guindani M, Leonardi M. Intraforaminal O(2)-O(3) versus periradicular steroidal infiltrations in lower back pain: randomized controlled study. AJNR Am J Neuroradiol. 2005 May;26(5):996-1000. PMID 15891150
- [Background] Bocci V, Luzzi E, Corradeschi F, Paulesu L, Di Stefano A. Studies on the biological effects of ozone: 3. An attempt to define conditions for optimal induction of cytokines. Lymphokine Cytokine Res. 1993 Apr;12(2):121-6. PMID 8324077
- [Background] Gibson JN, Grant IC, Waddell G. The Cochrane review of surgery for lumbar disc prolapse and degenerative lumbar spondylosis. Spine (Phila Pa 1976). 1999 Sep 1;24(17):1820-32. doi: 10.1097/00007632-199909010-00012. PMID 10488513
- [Derived] Bisshopp S, Linertova R, Carames MA, Szolna A, Jorge IJ, Navarro M, Melchiorsen B, Rodriguez-Diaz B, Gonzalez-Martin JM, Clavo B. Pain Relief, Disability, and Hospital Costs After Intradiscal Ozone Treatment or Microdiscectomy for Lumbar Disc Herniation: A 24-Month Real-World Prospective Study. J Clin Med. 2025 Jun 26;14(13):4534. doi: 10.3390/jcm14134534. PMID 40648907